CLINICAL TRIAL: NCT01264822
Title: Prognostic Study of Gastric MALT Lymphoma After Eradication of Helicobacter Pylori
Status: Completed | Type: Observational
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Other Study IDs: PRT10T
Record Dates: First submitted 2010-12-20; First posted 2010-12-22 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-01

CONDITIONS: Gastric Low-grade MALT Lymphoma With Helicobacter Pylori Positive
Keywords: Rabeprazole Sodium; Helicobacter pylori; stomach neoplasms
MeSH Terms: conditions — Stomach Neoplasms | interventions — Rabeprazole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Treatment Arm 1 Rabeprazole Sodium
  Interventions: Drug: Rabeprazole Sodium

INTERVENTIONS:
Drug: Rabeprazole Sodium — The following 3 drugs are taken orally at the same time twice daily for 7 days: rabeprazole sodium 10 mg, amoxicillin hydrate 750 mg, and clarithromycin 200 mg.
  The dose of clarithromycin may be properly increased as needed, although the upper limit is 400 mg twice daily.
  If Helicobacter pylori eradication with proton pump inhibitor, amoxicillin, and clarithromycin fails, the following 3 drugs will be taken at the same time twice daily for 7 days as an alternative treatment for adults: rabeprazole sodium 10 mg, amoxicillin hydrate 750 mg, and metronidazole 250 mg.

SUMMARY:
To survey the grade of gastric MALT lymphoma after eradication of Helicobacter pylori

ELIGIBILITY:
Inclusion criteria:

* gastric low-grade mucosa-associated lymphoid tissue (MALT) lymphoma with Helicobacter pylori positive
* The stages of MALT lymphoma are Lugano International Conference classification Stage I or II 1 and Wotherspoon grade 4 or 5

Exclusion criteria:

* With diffuse large B-cell lymphoma
* Have been treated to gastric mucosa-associated lymphoid tissue (MALT) lymphoma
* Corresponding to contraindication of each drug

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospitals and Clinics in Japan
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2011-01-13 (Actual); Primary Completion 2016-02-29 (Actual); Study Completion 2016-11-17 (Actual)

PRIMARY OUTCOMES:
Response rate of gastric low-grade MALT lymphoma by eradication of Helicobacter pylori | Every 3 months within the 1st year and every 6 months
Transition rate to secondary therapy for eradication of Helicobacter pylori | Every 6 months within the 1st year and every 12 months as needed

CONTACTS AND LOCATIONS:
Overall Officials: Katsuya Sugizaki, Study Director — Drug Fostering and Evolution Coordination Department, Eisai Co., Ltd.
Locations (42):
- Japan (42):
  - Nagoya, Aichi-ken
  - Hirosaki, Aomori
  - Kashiwa, Chiba
  - Matsuyama, Ehime
  - Fukuoka, Fukuoka
  - Fukuyama, Hiroshima
  - Hiroshima, Hiroshima
  - Sapporo, Hokkaido
  - Amagasaki-shi, Hyōgo
  - Kobe, Hyōgo
  - Hitachi, Ibaraki
  - Takamatsu, Kagawa-ken
  - Isehara, Kanagawa
  - Kyoto, Kyoto
  - Sendai, Miyagi
  - Nagano, Nagano
  - Suzaka, Nagano
  - Nagasaki, Nagasaki
  - Nara, Nara
  - Niigata, Niigata
  - Ōita, Oita Prefecture
  - Yufu, Oita Prefecture
  - Kurashiki, Okayama-ken
  - Okayama, Okayama-ken
  - Tsuyama, Okayama-ken
  - Hirakata, Osaka
  - Osaka, Osaka
  - Sayama, Osaka
  - Takatsuki, Osaka
  - Saga, Saga-ken
  - Matsue, Shimane
  - Hamamatsu, Shizuoka
  - Otawara-shi, Tochigi
  - Chūō, Tokyo
  - Minato-ku, Tokyo
  - Shinagawa-ku, Tokyo
  - tabashi City, Tokyo
  - Tottori-shi, Tottori
  - Toyama, Toyama
  - Yamagata, Yamagata
  - Ube, Yamaguchi
  - Yamaguchi, Yamaguchi